CLINICAL TRIAL: NCT04628312
Title: Standing Plantar Pressure Changes After Plantar Dry Needling in Flexor Digitorum Brevis
Brief Title: Foot Plantar Pressure Changes After Plantar Dry Needling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Head of Podiatry, Principal Investigator, and Physiotherapist, Mayuben Private Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2706201911419 C
Record Dates: First submitted 2020-11-07; First posted 2020-11-13 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Myofascial Pain Syndrome; Foot Diseases
MeSH Terms: conditions — Myofascial Pain Syndromes; Foot Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bilateral dry needling in Flexor Brevis Digitorum in subjects with latent trigger point (Experimental): Bilateral dry needling in Flexor Brevis Digitorum in subjects with latent trigger point
  Interventions: Other: Static footprint

INTERVENTIONS:
Other: Static footprint — The static footprint will measure the plantar pressures and surface area of the back of the foot, midfoot and forefoot. Subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned 30 degrees from the midline.

SUMMARY:
The aim of this clinical trial is to check the effects of dry needling in the Flexor digitorum Brevis.

Twenty healthy subjects wil be recruited for a quasi-experimental study. Participants will be from 18 to 40 years old, not obese. Participants will be measured before and after bilateral dry neddling in Flexor digitorum Brevis. The investigators will measure static footprint variables. The footprint variables will be divided in bilateral rear foot, bilateral midfoot, bilateral fore foot.

ELIGIBILITY:
Inclusion Criteria:

* Flat foot grade II or II with
* Must have latent trigger point in Flexor Brevis Digitorum muscles

Exclusion Criteria:

* Previous lower extremities surgery.
* History of lower extremities injury with residual symptoms (pain, "giving-away" sensations) within the last year.
* Leg-length discrepancy more than 1 cm

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Variables of plantar pressures with platform before dry puncture | Through study completion, an average of 1 week
  During 30 seconds we will record the plantar pressure variables in grams per square centimeter.
Variable footprint plantar surface with platform before dry puncture | Through study completion, an average of 1 week
  For 30 seconds we will record the area of the footprint in square centimeters.
Variables of plantar pressures with platform after dry puncture | Through study completion, an average of 1 week
  During 30 seconds we will record the plantar pressure variables in grams per square centimeter.
Variable footprint plantar surface with platform after dry puncture | Through study completion, an average of 1 week
  For 30 seconds we will record the area of the footprint in square centimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayuben Clinic, San Sebastián de los Reyes, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided